CLINICAL TRIAL: NCT07062679
Title: Effectiveness of Maitland Vs Mulligan Mobilization in Patient With Shoulder Pain
Brief Title: Maitland Vs Mulligan Mobilization in Patients With Shoulder Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC-01011 Shah Alam Khan
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Shoulder Pain
Keywords: Pain; Functional Status; Psychological Health Status
MeSH Terms: conditions — Shoulder Pain; Pain | interventions — Movement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Maitland Mobilization Oscillatory Glides
  Interventions: Other: Maitland Oscillatory Glides/Mobilization
- Group B (Experimental): Mulligan Mobilization with Movement (MWM)
  Interventions: Other: Mulligan Mobilization with Movement (MWM)

INTERVENTIONS:
Other: Maitland Oscillatory Glides/Mobilization — Hot pack for 15 minutes Ultrasound for 5 minutes Maitland Mobilization Oscillatory Glides inferiorly during normal abduction. Glenohumeral caudal glide mobilization was given at the rate of 2-3 glides per second for 30 seconds for each glide, 5 sets were given.
  (3 sessions per week for 4 weeks)
  Arms: Group A
Other: Mulligan Mobilization with Movement (MWM) — Hot pack for 15 minutes Ultrasound for 5 minutes Mobilization with Movement (MWM) Patient sitting with therapist posterolateral to him/her. Therapist places the Mulligan belt across the humeral head and to his waist. Patient movement (Flexion, extension, & abduction respectively) combined with therapist-applied joint gliding (postero-lateral Glide) MWM will be performed.
  3 sets of 10 reps per session (30 seconds rest between sets)
  (3 sessions per week for 4 weeks)
  Arms: Group B

SUMMARY:
* To find the effect of the Maitland Mobilization versus Mulligans Mobilization on the pain of the patient suffering from Shoulder pain.
* To determine the effectiveness of Mulligans Mobilization versus Maitland Mobilization on the functional status of the patient suffering from shoulder pain.
* To determine the effectiveness of Mulligans Mobilization versus Maitland Mobilization on the psychological health status of that patient.

DETAILED DESCRIPTION:
Shoulder is the most movable joint in the human body. A group of four muscles and their tendons, called the rotator cuff, give the shoulder its wide range of motion Rotator cuff muscles Swelling, damage, or bone changes around the rotator cuff can cause shoulder pain. Shoulder pain is highly prevalent and among musculoskeletal disorders is the third most common reason for visiting a primary care physician

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain from last 3 months to 1 year, Male and Female patients will be included & Age 20 years to 60 years.

Exclusion Criteria:

* Pain more than 1 year, Patients with certain shoulder structural deformities & Patients with autoimmune disease.

Ages: 3 Months to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Shoulder Pain Intensity Measured by Numeric Pain Rating Scale (NPRS) | 4 Weeks
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable") High test-retest reliability has been observed in both literate and illiterate patients with rheumatoid arthritis (r = 0.96 and 0.95, respectively) before and after medical consultation.
Shoulder Disability Level Measured by DASH (Disability of the Arm Shoulder and Hand Questionnaire) | 4 Weeks
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a 30-item questionnaire that looks at the ability of a patient to perform certain upper extremity activities.
Psychological Status Measured by Beck Depression Inventory Score | 4 Weeks
  The Beck Depression Inventory (BDI) is a 21-item questionnaire used to assess the severity of depressive symptoms. Scores range from 0 to 63, with higher scores indicating more severe symptoms. Interpretation of scores generally follows these guidelines: 0-13: minimal depression, 14-19: mild depression, 20-28: moderate depression, and 29-63: severe depression.
Cognitive & Emotional Response to Pain Measured by Pain Catastrophic Scale | 4 Weeks
  The Pain Catastrophizing Scale (PCS) is a 13-item self-report questionnaire that measures an individual's negative cognitive and emotional responses to pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Sadiq, MSPT (OMPT), Principal Investigator — Riphah International University
Locations (1):
- Saidu Group of Teaching Hospital Mingora Swat, Swāt, KPK, Pakistan